CLINICAL TRIAL: NCT05873491
Title: Homeless People in French-speaking Switzerland and Integrative Medicine: A Pilot Intervention in Music Therapy
Status: Completed | Type: Observational
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00514
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Homelessness
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Music therapy — The music therapy sessions will offer sensory workshops of immersive musical listening, digital and acoustic music creation and shared improvised music.

SUMMARY:
The goal of this observational study is to evaluate the feasibility to develop and implement a music therapy intervention among homeless individuals in French-speaking Switzerland.

The main questions it aims to answer are:

* Are the music therapy sessions acceptable?
* Are the music therapy sessions feasible?
* Are the chosen effectiveness primary outcomes appropriate for future larger studies (i.e., health-related quality of life and psychological stress)?

Participants will take part in six sub-group (of 6 participants) 2-hours music therapy sessions over 6 weeks. The sessions will be conducted by a certified music therapist and will offer sensory workshops of immersive musical listening, digital and acoustic music creation and shared improvised music. The music therapy sessions aim to create a space for sound and relaxation; promote the emergence of creativity and improvements in social skills and self-esteem through the co-construction of a privileged space for musical interaction.

DETAILED DESCRIPTION:
Study procedures:

The research team will recruit homeless service users within low-threshold institutions for homeless people in Lausanne and conduct the informed consent process. Participants agreeing to participate and providing written informed consent will complete a hetero-administrated paper-pencil questionnaire before receiving the first intervention session (T0). Parts of the dimensions assessed with this questionnaires (i.e., outcomes) will be reassessed after receiving the 6 music therapy sessions (T1).

At T0, the questionnaire will measure participants' demographics, health-related quality of life (QoL), psychological stress levels and self-esteem. Questionnaire completion will last between around 30 minutes each, depending on the support needed by the participants.

At T1, participants will complete a second questionnaire (T1). This questionnaire will assess the same dimensions than the ones at T0 except demographics and will also evaluate participants' satisfaction regarding the intervention sessions.

Quantitative assessment will be completed by qualitative evaluation through field observation during the 6 music therapy sessions by the research team. At T1, trained research staff will conduct one-on-one semi-structured interviews with the participants as well as with the music therapist. This qualitative assessment will aim at exploring therapist and participants' experience of the music therapy sessions. The semi-structured interview will last 30-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 ;
* Being fluent in French;
* Planning to stay in Lausanne the next 6 weeks;
* Committing to take part in as many as possible of the music therapy sessions;
* Agreeing to participate in group session;
* Being homeless according to the categories 1, 2, 3, or 5 of the ethos-light typology (Baptista & Marilier, 2019):

Living rough (i.e., public spaces); In emergency accommodation (i.e., overnight shelters); Living in accommodation for the homeless (i.e., temporary accommodation); Living in non-conventional dwellings due to lack of housing (i.e., mobile homes; non-conventional buildings);

Exclusion Criteria:

* Being unable to provide an informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include homeless adults in French-speaking Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-07-09 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Music therapy acceptability | week 1
  Acceptability will be measured based on the recruitment level (#included participants/#invited individuals). Specifically, we will monitor the number of participants invited to participate in the study and the acceptability outcome will be computed by dividing the number of participants who were included in the study by the number of participants who were invited to participate in the study.
Music therapy feasibility | week 1, week 2, week 3, week 4, week 5, week 6
  Feasibility will be measured based on participants' sessions participation level (#attended session/#total sessions). Specifically, we will monitor music therapy sessions attendance at week 1, 2, 3, 4, 5 and 6 for each included participants and the feasibility outcome will be computed by dividing the number of attended sessions by the total number of offered sessions (i.e., 6).

SECONDARY OUTCOMES:
Appropriateness of psychological distress outcome for future clinical trials | week 1 and week 6
  In line with similar past pilot research among homeless individuals (Gaddy, 2018; Garland et al., 2016; Maddock et al., 2017), this questionnaire will evaluate psychological distress with the Kessler Psychological Distress Scale (K6) (Furukawa et al., 2003).
Appropriateness of quality of life outcome for future clinical trials | week 1 and week 6
  Perceived QoL using the World Health Organization Quality of Life-BREF (Skevington et al., 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Véronique S Grazioli, PhD, Principal Investigator — Center for Primary Care and Public Health
Locations (1):
- Center for Primary Care and Public Health, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
For confidentiality issues and due to the small sample planned in this feasibility pilot study, we do not plan to share data.

REFERENCES:
- [Background] Gaddy MA. Implementation of an integrative medicine treatment program at a Veterans Health Administration residential mental health facility. Psychol Serv. 2018 Nov;15(4):503-509. doi: 10.1037/ser0000189. Epub 2017 Oct 12. PMID 29022737
- [Background] Maddock, A., D. Hevey, and K. Eidenmuller, Mindfulness training as a clinical intervention with homeless adults: A pilot study. International Journal of Mental Health Addiction, 2017. 15: p. 529-544.
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Furukawa TA, Kessler RC, Slade T, Andrews G. The performance of the K6 and K10 screening scales for psychological distress in the Australian National Survey of Mental Health and Well-Being. Psychol Med. 2003 Feb;33(2):357-62. doi: 10.1017/s0033291702006700. PMID 12622315
- [Background] Baptista, I. and E. Marilier, Fighting homelessness and housing exclusion in Europe: A study of national policies, E.S.P.N. (ESPN), Editor. 2019: Brussels: European Commission.
- [Background] Garland EL, Roberts-Lewis A, Tronnier CD, Graves R, Kelley K. Mindfulness-Oriented Recovery Enhancement versus CBT for co-occurring substance dependence, traumatic stress, and psychiatric disorders: Proximal outcomes from a pragmatic randomized trial. Behav Res Ther. 2016 Feb;77:7-16. doi: 10.1016/j.brat.2015.11.012. Epub 2015 Nov 27. PMID 26701171